CLINICAL TRIAL: NCT00293618
Title: IMplementation of a Prediction Rule in Anesthesia Practice to Improve Cost-Effectiveness of Treatment of Postoperative Nausea and Vomiting
Brief Title: Implementation Study of the PostOperative Nausea and Vomiting Prediction Rule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: K.G.M.Moons, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05/288; 945-16-202
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Implementation of prediction rules; Decision Support Systems, Clinical; PONV; Emesis; Nausea; Vomiting; Postoperative; Implementation; prediction rule; impact study; decision support; clinical decision support
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting; Nausea | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Arm of anesthesiologists and senior residents who receive a patient's individual predicted PONV risk intraoperatively
  Interventions: Device: Automatic Risk Presentation in the operating room; Other: Education; Other: Feedback
- Usual Care (Active Comparator): Anesthesiologists and senior residents who provide usual care: they provide PONV prophylaxis as they always have
  Interventions: Other: Education

INTERVENTIONS:
Device: Automatic Risk Presentation in the operating room — Automatic calculation and presentation of a patient's individual predicted PONV risk by the anesthesia information management system during the entire procedure
  Arms: Intervention
Other: Education — Specific information is provided to the intervention group: about PONV, about the prediction model. While the Usual Care group only receives information about the study purposes
Other: Feedback — Feedback about the physician's personal performance on prevention of PONV
  Arms: Intervention

SUMMARY:
This study evaluates whether the implementation of a prediction rule for postoperative nausea and vomiting changes physician behaviour, improves patient outcome and improves cost-effectiveness of treatment of postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Background and objectives. So-called prediction rules (risk scores) have become increasingly popular in all medical disciplines. This will only rise with the introduction of electronic patient records as these will enhance their use. However, effects of implementation of such rules in daily care has hardly been studied. Also not in anesthesiology. We developed and validated an accurate rule to preoperatively predict the risk of postoperative nausea and vomiting (PONV) in surgical inpatients. PONV causes extreme patient discomfort and occurs in even 30%-50% of all surgical inpatients. As routine administration of PONV prophylaxis is not cost-effective, a risk-tailored approach using an accurate prediction rule is widely advocated. Before large-scale implementation, we aim to study whether such implementation indeed changes physician behavior and improves patient outcome. Given the increase interest in prediction rules, another aim is to study general causes of successful/poor implementation of prediction rules in health care. Design. Cluster, randomized study in which 60 anesthesiologists and senior residents of the UMC Utrecht will be randomized to either the intervention or usual care group.

Study population. Adult,elective,non-ambulatory,surgical patients undergoing general anesthesia of UMC Utrecht.

Intervention. Implementation of risk-tailored PONV strategy (use of the PONV prediction rule with suggested anti-emetic strategies per risk group) in current care.

Outcomes. Primary:incidence of PONV in first 24 hours. Secondary:change in anesthesiologists' behavior in terms of administered anti-emetic management, cost-effectiveness of intervention, attitudes of physicians towards prediction rules in general.

Sample size. 11,000

Economic evaluation. Estimation of incremental costs per prevented PONV case.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Undergoing elective surgery
* General anesthesia

Exclusion Criteria:

* emergency surgery
* postoperative transfer to ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11970 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
the incidence of PONV within the first 24 hours | within 24 hours after surgery

SECONDARY OUTCOMES:
Behaviour of the anaesthesiologist regarding PONV-prophylaxis | Perioperative
Cost-effectiveness risk-based prophylaxis compared to standard care | Within 24 hours after surgery
Attitude of anesthesiologists to use risk estimations from a prediction rule | At the start and end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Cor J Kalkman, M.D. PhD, Study Chair — UMC Utrecht; Karel G Moons, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Kappen TH, Moons KG, van Wolfswinkel L, Kalkman CJ, Vergouwe Y, van Klei WA. Impact of risk assessments on prophylactic antiemetic prescription and the incidence of postoperative nausea and vomiting: a cluster-randomized trial. Anesthesiology. 2014 Feb;120(2):343-54. doi: 10.1097/ALN.0000000000000009. PMID 24105403
- [Derived] van Dijk JF, Kappen TH, van Wijck AJ, Kalkman CJ, Schuurmans MJ. The diagnostic value of the numeric pain rating scale in older postoperative patients. J Clin Nurs. 2012 Nov;21(21-22):3018-24. doi: 10.1111/j.1365-2702.2012.04288.x. PMID 23083383
- [Derived] van Dijk JF, van Wijck AJ, Kappen TH, Peelen LM, Kalkman CJ, Schuurmans MJ. Postoperative pain assessment based on numeric ratings is not the same for patients and professionals: a cross-sectional study. Int J Nurs Stud. 2012 Jan;49(1):65-71. doi: 10.1016/j.ijnurstu.2011.07.009. Epub 2011 Aug 15. PMID 21840522